CLINICAL TRIAL: NCT00319865
Title: PS-341 (Bortezomib, Velcade®), Adriamycin and Dexamethasone (PAD) Combination Therapy Followed by Thalidomide With Dexamethasone (Thal/Dex) for Relapsed or Refractory Multiple Myeloma
Brief Title: PAD Combination Therapy Followed by Thal/Dex for Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Multiple Myeloma Working Party (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMM55
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma Relapsed
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide; Doxorubicin; Dexamethasone

INTERVENTIONS:
Drug: Velcade
Drug: Thalidomide
Drug: Adriamycin
Drug: Dexamethasone

SUMMARY:
Prospective multicenter phase 2 study using PAD and Thal/Dex combination sequentially.

DETAILED DESCRIPTION:
Although the overall survival was improved with the introduction of high dose therapy with autologous hematopoetic stem cell transplantation,it remains as a incurable disease. Most patients ultimately relapse. Recenlty, targeted therapy using novel agents, such as bortezomib and thalidomide, shows the possibility of improved in this situation. Among them, PAD (Velcade, Adriamycin,Dexamethasone) showed highest response rate. PAD does not show any cross resiatance with another effective combination, thalidomide plus dexamethasone.

We desined prospective multicenter phase 2 study using these combination sequentially.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who relapsed after at least 1 lines of therapy including high dose thearapy with autologous stem cell transplantation and chemotherapy.
* Presence of measureble disease : serum M-protein > 1g/dL or urine M-protein > 400mg/day
* Age < 75
* Performance status </= ECOG 2
* Expected survival > 6 months
* who signs the informed consent

Exclusion Criteria:

* known hypersensitivity to thalidomide or dexamethasone
* known refractoriness to thalidomide + dexamethasone
* Previous Velcade therapy
* Sepsis
* Woman in reproductive age
* Serum creatinine > 2 mg/dL ; 24 hour creatinine clearance < 30 ml/min; past medical history of kidney transplatation
* Peripheral neuropathy >/= grade 2
* Recurrent DVT or pulmonary embolism
* Cardiac ejection fraction <0.5 : Severe conduction disorder
* Hepatic dysfunction (AST or ALT ≥ x 5 upper normal) or active hepatitis
* Active ulcers in gastrofiberscope

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47
Dates: Start 2005-11; Study Completion 2008-09

PRIMARY OUTCOMES:
Response rate of PAD induction Therapy

SECONDARY OUTCOMES:
Response rate of PAD followed by Thal/Dex maintenance
Progression free survival and Overall survival of PAD/Thal-Dex.
To evaluate toxicities of PAD/Thal-Dex

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hoon Lee, M.D., Principal Investigator — Korean Multiple Myeloma Working Party
Locations (1):
- Gachon University Gil Hospital, Inchon, South Korea

REFERENCES:
- See also: Korean Society of Hematology — http://www.hematology.or.kr/